CLINICAL TRIAL: NCT00999791
Title: Intravitreal Diclofenac Versus Avastin as Primary Treatment of Diffuse Diabetic Macular Edema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Model: Parallel | Purpose: Treatment
Other Study IDs: 8818
Record Dates: First submitted 2009-07-07; First posted 2009-10-22 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-10

CONDITIONS: Diffuse Diabetic Macular Edema
MeSH Terms: interventions — Bevacizumab; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avastin (Active Comparator)
  Interventions: Drug: Bevacizumab
- Diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Bevacizumab
  Arms: Avastin
Drug: Diclofenac
  Arms: Diclofenac

SUMMARY:
Diffuse Macular Edema is the main cause of visual disorders in diabetic patients.

Diclofenac is a cheap drug available in most of treatment centers.in animal studies the safe dosage is identified that can be used in diffuse diabetic macular edema for treatment. in this study, we are going to compare the effect of intra vitreal injection of Diclofenac and Bevacizumab in primary treatment of diffuse diabetic macular edema.

DETAILED DESCRIPTION:
Diffuse Macular Edema is the main cause of visual disorders in diabetic patients.

Diclofenac is a cheap drug available in most of treatment centers.in animal studies the safe dosage is identified that can be used in diffuse diabetic macular edema for treatment. in this study, we are going to compare the effect of intra vitreal injection of Diclofenac and Bevacizumab in primary treatment of diffuse diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically significant macular edema and diffuse macular edema

Exclusion Criteria:

* any history of focal photocoagulation
* any prior intra ocular injection
* history of glaucoma with high pressure
* history of ophthalmic surgery
* high rish PDR
* active PDR

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2009-07

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran